CLINICAL TRIAL: NCT02098564
Title: The Effect of Activity-based Training in Patients With Hand-related Injuries Grouped Using Sense of Coherence Scores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Region of Southern Denmark (Other); Bevica Fonden (Other); Danish Association of Occupational Therapist (Other)
Responsible Party: Principal Investigator, Alice Ørts Hansen, OT, Master in health science, Ph.D. student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REHAB123
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hand Related Injuries
Keywords: hand therapy; activity-based training; hand related injuries; sense of coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- strong sense of coherence control group (Active Comparator): Patients with a strong sense of coherence. Participants will perform joint mobility exercises which are appropriate for their injury, both in the therapy setting and as a home exercise program.
  Interventions: Other: Joint mobility exercises hand therapy
- strong sense of coherence intervention (Experimental): Patients with a strong sense of coherence. Participants will perform joint mobility exercises which are appropriate for their injury and specific meaningful activities which they performed prior to the hand-related injury. This will be performed both in the therapy setting and as a home exercise program.
  Interventions: Other: activity-based hand therapy
- weak sense of coherence control group (Active Comparator): Patients with a weak sense of coherence. Participants will perform joint mobility exercises which are appropriate for their injury, both in the therapy setting and as a home exercise program.
  Interventions: Other: Joint mobility exercises hand therapy
- weak sense of coherence intervention (Experimental): Patients with a weak sense of coherence. Participants will perform joint mobility exercises which are appropriate for their injury and specific meaningful activities which they performed prior to the hand-related injury. This will be performed both in the therapy setting and as a home exercise program.
  Interventions: Other: activity-based hand therapy
- medium sense of coherence intervention (Experimental): Patients with a medium sense of coherence. Participants will perform joint mobility exercises which are appropriate for their injury and specific meaningful activities which they performed prior to the hand-related injury. This will be performed both in the therapy setting and as a home exercise program.
  Interventions: Other: activity-based hand therapy
- medium sense of coherence control group (Active Comparator): Patients with a weak sense of coherence. Participants will perform joint mobility exercises which are appropriate for their injury, both in the therapy setting and as a home exercise program.
  Interventions: Other: Joint mobility exercises hand therapy

INTERVENTIONS:
Other: Joint mobility exercises hand therapy — Joint mobility exercises which are appropriate for their injury, both in the therapy setting and as a home exercise program
  Arms: medium sense of coherence control group; strong sense of coherence control group; weak sense of coherence control group
Other: activity-based hand therapy — intervention involve joint mobility exercises which are appropriate for their injury and training with specific meaningful activities which they performed prior to the hand-related injury. Activity-based hand therapy will be performed both in the therapy setting and as a home exercise program.
  Arms: medium sense of coherence intervention; strong sense of coherence intervention; weak sense of coherence intervention

SUMMARY:
Background Patients with the same type of hand injury often reach different functional levels. Therefore, it is necessary to investigate what kind of rehabilitation is most efficient for each individual patient.

Research has shown that a person's "Sense of Coherence" (SOC) affects how he /she deals with disease. Furthermore, SOC can help predict final outcomes after orthopedic injuries and should therefore; be taken into consideration when planning rehabilitation. It was concluded in a study that patients with a weak SOC who have had a hand injury, may benefit from extra support to manage their everyday activities in order to reach the same final outcome as patients with a strong SOC.

Purpose To investigate two types of rehabilitation on patients with a hand-related injury (joint mobility exercises vs. activity-based training and joint mobility exercises) and to investigate whether SOC can be used as an indicator of which patients would benefit from activity-based training.

Hypotheses

1. Patients with a hand-related injury will benefit from activity-based training in their rehabilitation program.
2. Patients with a weak SOC will achieve the best functional level, if activity-based training is included in their rehabilitation program.
3. Patients with a strong SOC will not achieve a higher functional level, if activity-based training is included in their rehabilitation program.

Study design Randomised control trial. Methods Four-hundred-twenty- patients age 18 years or older are included when referred to specialized outpatient occupational therapy after a hand-related injury. To ensure sufficient and balanced patient variation in relation to pre-rehabilitation sense of coherence, a balanced randomisation principle has been implemented.

Data will be collected through questionnaires. The questionnaires measure SOC (13 items version), function (DASH), quality of life (EQ5D) and satisfaction.

All participants will perform joint mobility exercises which are appropriate for their injury. In addition, participants who will be performing activity-based training will train with specific meaningful activities which they performed prior to the hand-related injury.

Clinical relevance The knowledge obtained will be incorporated into the planning of occupational therapy rehabilitation services for this patient group, so that the patients will receive the most optimal conditions in which to achieve their previous level of function after a hand injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hand-related diagnoses (acute injuries or elective surgeries)
* Patients referred to specialized outpatient occupational therapy rehabilitation at Odense University Hospital
* Patients who are able to understand, speak and read enough Danish to participate
* 18-years of age or older

Exclusion Criteria:

* A rehabilitation treatment period under four weeks and less than three treatments
* Dementia or cognitive impairments
* Where it is not considered medically or therapeutically safe to allow the patient to be included in the randomization process.
* Patients with shoulder problems
* Patients with epicondylitis
* Patients with plexus brachialis injuries
* Patients who only have difficulty extending their non-dominant 5th finger.
* Burn injuries
* Pt. who have had a CMP joint replacement operation because of arthrosis (Swanson)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand questionnaire | from baseline to 12 months after start of rehabilitation

SECONDARY OUTCOMES:
The EQ-5D Quality of life questionnaire | From baseline to 3 months
Sense of Coherence Questionnaire | From baseline to 12 months
  13 items questionnaire
Canadian Occupational Performance Measure (COPM) Canadian Occupational Performance Measure (COPM) | From baseline to 3 months
Satisfaction with daily living and rehabilitation | From baseline to12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans B Tromborg, Ph.D, Study Chair — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark